CLINICAL TRIAL: NCT02632955
Title: Drug Eluting Balloon for Early Fistula Failure Trial
Acronym: DEBEFF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Naveed Ul Haq, Director of Dialysis Access & Interventional Nephrology Program, King Faisal Specialist Hospital & Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2151 054
Record Dates: First submitted 2015-12-15; First posted 2015-12-17 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Stenosis of Arteriovenous Dialysis Fistula
Keywords: arteriovenous fistula; hemodialysis; drug coated balloon
MeSH Terms: conditions — Arteriovenous Fistula | interventions — Angioplasty, Balloon, Coronary

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug Eluting Balloon (Experimental): After pre dilation of the lesion with regular angioplasty balloon, drug coated balloon Lutonix(R) by Bard Inc. will be introduced over the lesion as quickly as possible. Lutonix is a paclitaxel coated balloon which delivers the drug locally. The diameter of the drug coated balloon will be same as the diameter of the largest balloon used for pre dilation. Drug coated balloon will be inflated not exceeding the rated burst pressure. The minimum inflation time will be 1 minute.
  Interventions: Drug: Drug Eluting Balloon
- Regular Angioplasty (Sham Comparator): After predilation of the lesion with regular balloon, the same balloon will be reintroduced without the drug to be inflated for a minimum of 1 minute. This angioplasty will not deliver any local drug.
  Interventions: Procedure: Regular angioplasty

INTERVENTIONS:
Drug: Drug Eluting Balloon — After pre dilation of the lesion with regular angioplasty balloon, drug coated balloon Lutonix(R) by Bard Inc. will be introduced over the lesion as quickly as possible. Lutonix is a paclitaxel coated balloon which delivers the drug locally. The diameter of the drug coated balloon will be same as the diameter of the largest balloon used for pre dilation. Drug coated balloon will be inflated not exceeding the rated burst pressure. The minimum inflation time will be 1 minute.
  Other Names: Lutonix drug eluting Balloon angioplasty
  Arms: Drug Eluting Balloon
Procedure: Regular angioplasty — After predilation of the lesion with regular balloon, the same balloon will be reintroduced without the drug to be inflated for a minimum of 1 minute. This angioplasty will not deliver any local drug.
  Other Names: Percutaneous balloon angioplasty
  Arms: Regular Angioplasty

SUMMARY:
Hemodialysis (HD) remains the most prevalent form of renal replacement therapy (RRT) for patients with End Stage Renal Disease (ESRD). Loss and dysfunction of vascular access is a significant contributor to morbidity in ESRD patients on HD. The National Kidney Foundation's Kidney Disease Outcomes Quality Initiative (KDOQI) guidelines suggest that all ESRD patients should initiate dialysis with a functioning permanent vascular access with arteriovenous fistulas (AVF) preferred over arteriovenous grafts (AVG). Central venous catheters (CVC) are the least preferred vascular access for HD due to the complications associated with them. Despite these recommendations, up to 80% patients start dialysis with a CVC. One of the reasons for low AVF rates is early fistula failure (EFF). The most important causes for EFF amenable to intervention is stenosis anywhere in the circuit. Endovascular approach has shown a high rate of technical success in the treatment of stenotic lesions related to HD arteriovenous access. Percutaneous balloon angioplasty (PBA) is considered the treatment of choice for these lesions. Despite good technical and immediate success PBA has poor long term outcomes with recurrence rates of 60-70% at 6 months. One of the reasons could be the damage caused by angioplasty itself leading to intima-media rupture promoting the cascade of events leading to further development of neo intimal hyperplasia (NIH). Recently the use of covered stents at the time of angioplasty has shown better patency rates at 6 months but still not optimal. Lately the development of drug eluting stents and drug eluting balloons (DEB) have shown considerable advantage in clinical trials related to coronary and peripheral arterial disease angioplasty. In a randomized control trial, the researchers are planning to assess the efficacy of DEB angioplasty as compared to standard PBA in AVF's with EFF.

DETAILED DESCRIPTION:
Hemodialysis (HD) remains the most prevalent form of RRT for patients with End Stage Renal Disease (ESRD). Just in the United States there are more than 380,000 patients with ESRD on hemodialysis (HD) and the number is expected to increase to 500,000 by the year 2020. Recent data provided by Saudi Centre for Organ Transplantation (www.scot.org.sa) shows that there are just over 13000 patients with End-stage renal disease (ESRD) on hemodialysis in the Kingdom of Saudi Arabia. This number is expected to rise at a rate of 7-8% annually reaching 18000 by year 2018. Establishing a viable vascular access is crucial and is considered the 'life-line' for such patients. Loss and dysfunction of vascular access is a significant contributor to morbidity in ESRD patients on HD. In the United States <50% of all hemodialysis accesses remain patent at 3 years with the economic burden of maintaining vascular access patency calculated to exceed $1 billion with a >6% annual trend. The National Kidney Foundation's Kidney Disease Outcomes Quality Initiative (KDOQI) guidelines suggest that all ESRD patients should initiate dialysis with a functioning permanent vascular access with arteriovenous fistulas (AVF) preferred over arteriovenous grafts (AVG). Central venous catheters (CVC) are the least preferred vascular access for HD due to the complications associated with them. Despite these recommendations and clear benefits of using arteriovenous access for hemodialysis, up to 80% patients start dialysis with a CVC. One of the reasons for low AVF rates is early fistula failure (EFF). EFF is defined as an AVF that never develops adequately for dialysis (failure to mature) or which fails within 3 months of starting dialysis. An adequate AVF for dialysis according to KDOQI guidelines is the one which a) Has a flow of greater than 600ml/min, b) Has a diameter of 0.6cm or greater and c) Is approximately not deeper than 0.6cm from the skin surface. Between 23%-46% of newly constructed AVF have problems with early failure resulting in a dismal one year patency of 60-65%.

In order to devise a strategy to prevent EFF, one needs to understand the physiology of fistula maturation. Creation of an AVF leads to an immediate increase in flow through the vein due to the pressure gradient created. This increase in flow leads to increase wall shear stress which is defined mathematically by the formula 4ηQ/πr3, where η is blood viscosity, Q is blood flow and r is vessel radius. Shear stress thus is directly proportional to blood flow while inversely proportional to vessel diameter. After the creation of the AVF, the flow mediated increase in shear stress is mitigated by vessel dilatation through biological mediators. Consequently the shear stress is brought back to pre-anastomosis levels leading to vessel dilation. It seems that this positive remodeling of the vein leading to AVF maturation is dependent on increase in blood flow rather than the increase in pressure. Any pathology affecting the blood flow through the newly constructed AVF can thus lead to failure to mature.

The two most important causes for EFF amenable to intervention are stenosis anywhere in the circuit (present in around 80% of EFF) and/or presence of accessory veins. While stenosis development is pathological and accessory vein presence is natural, both lead to decreased blood flow through the main AVF circuit, which may be responsible for failure to mature. Addressing these two entities in a timely fashion can lead to salvage of many AVF, which otherwise would have been abandoned.

Development of neo-intimal hyperplasia (NIH) is the main pathology causing stenosis in the AVF circuit. There are many factors thought to be responsible for the development of this NIH. These include turbulent flow with wall shear stress disturbances, uremic endothelial dysfunction, repeated venipunctures, and unique anatomic factors. The pathogenesis includes migration of smooth muscle cells and myofibroblasts from media to intima, neoangiogenesis of microvessels inside neointima, and high levels of inflammatory blood markers.

Since its introduction, endovascular approach has shown a high rate of technical success in the treatment of stenotic lesions related to HD arteriovenous access. Percutaneous balloon angioplasty (PBA) is considered the treatment of choice for these lesions. Despite good technical and immediate success PBA has poor long term outcomes with recurrence rates of 60-70% at 6 months. One of the reasons could be the damage caused by angioplasty itself leading to intima-media rupture promoting the cascade of events leading to further development of NIH. Recently the use of covered stents at the time of angioplasty has shown better patency rates at 6 months but still not optimal. Lately the idea of delivering loco-regional pharmacological agents at the time of angioplasty to prevent NIH from happening has been extensively studied mostly in coronary arteries. This lead to the development of drug eluting stents and drug eluting balloons (DEB). These therapies have shown considerable advantage in clinical trials related to coronary and peripheral arterial disease. Although promising but advantages in coronary and peripheral arteries may not be applicable to arteriovenous access where the lesions are mostly venous with different characteristics. The role of these more costly interventions needs to be addressed in stenosis related to AVF, before wide spread use can be recommended. In a recent randomized non-blinded study involving 40 patients, Kostanos et al showed better 6 month patency rates (70% vs 25%) with DEB angioplasty as compared to standard PBA. The study is non-blinded and involved both AVG and AVF with target lesion spread all over the arteriovenous access circuit. Patane et al recently performed a study on 26 failing radiocephalic AVF's with juxta-anastamosis stenosis, defined as stenosis within 3 cm of arteriovenous anastamosis. In this study DEB angioplasty showed a 6 month primary patency of 96.1% which is much higher than historical conventional balloon angioplasty. The investigators targeted a lesion which resembles more closely arterial lesions where DEB has been shown to be effective, which seems more reasonable but there were no controls in the study. Due to the lack of a control group such high patency rates become questionable. Nevertheless this study highlights the importance of doing a randomized control trial targeting a specific lesion. In a controlled pilot study of radio-cephalic AVF with inflow stenosis Lai et al from Taiwan showed short term patency benefits with DEB angioplasty as compared to standard PBA. This being a pilot study had only 20 patients and was not adequately powered to answer the question. If these results are indeed proven to be true, this can lead to great improvement in patency of AVF's. In a randomized control trial the researchers are planning to assess the efficacy of DEB angioplasty as compared to standard PBA in AVF's with EFF.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Patients with EFF
* Stenosis anywhere in the AVF being the only identifiable cause of EFF.

Exclusion Criteria:

* Patients with AVF which is deeper than 0.8cm from the skin.
* AVF which is tortuous and lacks adequate straight segment for cannulation with 2 needles.
* Patients with allergy to paclitaxel
* Patients on anti-coagulation and those with bleeding disorders.
* Severe thrombocytopenia i.e platelet count< 50,000.
* Life expectancy less than 12 months.
* Documented severe contrast allergy.
* Inability to come for timely and adequate follow up.
* Patients undergoing transplantation work up and expected to be transplanted within 6 months.
* EFF secondary to accessory veins or causes other than stenosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Primary patency | 6 months
  Patency of AVF without any additional procedures. Patency is defined as supporting HD with a pump speed of at least 300ml/min.

SECONDARY OUTCOMES:
Secondary Patency | 6 months
  Patency of AVF with additional procedures.Patency is defined as supporting HD with a pump speed of at least 300ml/min.

CONTACTS AND LOCATIONS:
Overall Officials: Naveed U Haq, MD, FASN, Principal Investigator — King Faisal Specialist Hospital & Research Center
Locations (1):
- King Faisal Specialist Hospital & Research Center, Riyadh, Saudi Arabia

REFERENCES:
- [Background] Beathard GA, Arnold P, Jackson J, Litchfield T; Physician Operators Forum of RMS Lifeline. Aggressive treatment of early fistula failure. Kidney Int. 2003 Oct;64(4):1487-94. doi: 10.1046/j.1523-1755.2003.00210.x. PMID 12969170
- [Background] Roy-Chaudhury P, Spergel LM, Besarab A, Asif A, Ravani P. Biology of arteriovenous fistula failure. J Nephrol. 2007 Mar-Apr;20(2):150-63. PMID 17514619
- [Background] Beathard GA, Settle SM, Shields MW. Salvage of the nonfunctioning arteriovenous fistula. Am J Kidney Dis. 1999 May;33(5):910-6. doi: 10.1016/s0272-6386(99)70425-7. PMID 10213648
- [Background] Turmel-Rodrigues L, Mouton A, Birmele B, Billaux L, Ammar N, Grezard O, Hauss S, Pengloan J. Salvage of immature forearm fistulas for haemodialysis by interventional radiology. Nephrol Dial Transplant. 2001 Dec;16(12):2365-71. doi: 10.1093/ndt/16.12.2365. PMID 11733628
- [Background] Roy-Chaudhury P, Arend L, Zhang J, Krishnamoorthy M, Wang Y, Banerjee R, Samaha A, Munda R. Neointimal hyperplasia in early arteriovenous fistula failure. Am J Kidney Dis. 2007 Nov;50(5):782-90. doi: 10.1053/j.ajkd.2007.07.019. PMID 17954291
- [Background] Asif A, Lenz O, Merrill D, Cherla G, Cipleu CD, Ellis R, Francois B, Epstein DL, Pennell P. Percutaneous management of perianastomotic stenosis in arteriovenous fistulae: results of a prospective study. Kidney Int. 2006 May;69(10):1904-9. doi: 10.1038/sj.ki.5000358. PMID 16557220
- [Background] Haskal ZJ, Trerotola S, Dolmatch B, Schuman E, Altman S, Mietling S, Berman S, McLennan G, Trimmer C, Ross J, Vesely T. Stent graft versus balloon angioplasty for failing dialysis-access grafts. N Engl J Med. 2010 Feb 11;362(6):494-503. doi: 10.1056/NEJMoa0902045. PMID 20147715
- [Background] Stettler C, Wandel S, Allemann S, Kastrati A, Morice MC, Schomig A, Pfisterer ME, Stone GW, Leon MB, de Lezo JS, Goy JJ, Park SJ, Sabate M, Suttorp MJ, Kelbaek H, Spaulding C, Menichelli M, Vermeersch P, Dirksen MT, Cervinka P, Petronio AS, Nordmann AJ, Diem P, Meier B, Zwahlen M, Reichenbach S, Trelle S, Windecker S, Juni P. Outcomes associated with drug-eluting and bare-metal stents: a collaborative network meta-analysis. Lancet. 2007 Sep 15;370(9591):937-48. doi: 10.1016/S0140-6736(07)61444-5. PMID 17869634
- [Background] Cassese S, Byrne RA, Ott I, Ndrepepa G, Nerad M, Kastrati A, Fusaro M. Paclitaxel-coated versus uncoated balloon angioplasty reduces target lesion revascularization in patients with femoropopliteal arterial disease: a meta-analysis of randomized trials. Circ Cardiovasc Interv. 2012 Aug 1;5(4):582-9. doi: 10.1161/CIRCINTERVENTIONS.112.969972. Epub 2012 Jul 31. PMID 22851526
- [Background] Katsanos K, Karnabatidis D, Kitrou P, Spiliopoulos S, Christeas N, Siablis D. Paclitaxel-coated balloon angioplasty vs. plain balloon dilation for the treatment of failing dialysis access: 6-month interim results from a prospective randomized controlled trial. J Endovasc Ther. 2012 Apr;19(2):263-72. doi: 10.1583/11-3690.1. PMID 22545894
- [Background] Patane D, Giuffrida S, Morale W, L'Anfusa G, Puliatti D, Bisceglie P, Seminara G, Calcara G, Di Landro D, Malfa P. Drug-eluting balloon for the treatment of failing hemodialytic radiocephalic arteriovenous fistulas: our experience in the treatment of juxta-anastomotic stenoses. J Vasc Access. 2014 Sep-Oct;15(5):338-43. doi: 10.5301/jva.5000211. Epub 2014 Feb 10. PMID 24531999
- [Background] Lai CC, Fang HC, Tseng CJ, Liu CP, Mar GY. Percutaneous angioplasty using a paclitaxel-coated balloon improves target lesion restenosis on inflow lesions of autogenous radiocephalic fistulas: a pilot study. J Vasc Interv Radiol. 2014 Apr;25(4):535-41. doi: 10.1016/j.jvir.2013.12.014. Epub 2014 Feb 12. PMID 24529550